CLINICAL TRIAL: NCT02126397
Title: Comparative Study of Endometrial Polypectomy Performed With Bipolar Electrode Versapoint and Laser Diode. A Randomised Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel Bejerano Blázquez (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Universidad Nacional de Córdoba (Other)
Responsible Party: Sponsor-Investigator, Isabel Bejerano Blázquez, IMIBIC, Maimónides Biomedical Research Institute of Córdoba
Organization: Maimónides Biomedical Research Institute of Córdoba (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 230485
Record Dates: First submitted 2014-01-28; First posted 2014-04-30 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Endometrial Polyps
Keywords: endometrial polyp; resection of endometrial polyps; hysteroscopy; bipolar electrode Versapoint; Laser Diode
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- polyps resection with Laser Diode (Active Comparator): application of the laser diode by hysteroscopy to remove the endometrial polyp
  Interventions: Procedure: polyps resection with Laser Diode
- polyps resection with bipolar electrode (Active Comparator): application of the bipolar electrode Versapoint by hysteroscopy to remove the endometrial polyp
  Interventions: Procedure: polyps resection with bipolar electrode

INTERVENTIONS:
Procedure: polyps resection with Laser Diode — resection of endometrial polyps by hysteroscopy without anesthesia
  Arms: polyps resection with Laser Diode
Procedure: polyps resection with bipolar electrode
  Arms: polyps resection with bipolar electrode

SUMMARY:
Hysteroscopy today is considered the gold standard for the diagnosis and treatment of endometrial polyps. In recent years we have used the bipolar energy for resection of polyps by hysteroscopy, becoming a routine clinical practice and universally accepted.

Resection of endometrial polyps laser energy has recently begun to be used with satisfactory results, so studies are needed to analyze these results and compare it with the usual techniques .

This time in advance of medicine, it is appropriate to introduce minimally invasive procedures , allowing resection of endometrial polyps on an outpatient basis without anesthesia and acceptable to most patients.

These procedures assume a lower cost and are associated with a lower surgical risk due to their realization without anesthesia .

Hypothesis: Resection of polyps outpatient laser diode has a similar or superior to that of the bipolar electrode tolerability. The diode laser is a viable , quick , simple technique with a high percentage of resection and high degree of satisfaction of patients

DETAILED DESCRIPTION:
Main objective: To assess the tolerability of diode laser in the treatment of endometrial polyps using a visual analogue pain scale.

Secondary objectives:

* Determine if complete resection of polyps is achieved with both methods.
* Compare the time spent on the removal of the polyp in each of the hysteroscopic methods.
* To evaluate the safety of the laser diode with respect to the bipolar electrode (vagal syndrome, uterine perforation, infection, bleeding).
* Assess the recurrence of polyps after 3 months of resection (via hysteroscopy).
* Compare the degree of patient satisfaction with the different methods.

Design: randomized single blind clinical trial corresponds to an experimental analytical study. The patients randomly into 2 groups will include: Group A bipolar electrode treatment Versapoint and Group B diode laser treatment. Randomization was performed using a random table with 2 groups, generated in Microsoft Office Excel. The sample size needed to detect a difference in visual analog pain scale of a point with respect to the laser diode bipolar electrode is calculated; assuming a standard deviation of 1.75, a sample size of 49 patients in each group (98 would be needed in total), to a level of significance of 5% (0.05 α) with a power of 0.80 (beta 0.20). Assuming a loss of individuals from 5 to 10%

ELIGIBILITY:
Inclusion Criteria:

* patients previously diagnosed of endometrial polyps that can be resected. The diagnosis will be made hysteroscopically. The patient must be informed about the study, and sign the informed consent.

Exclusion Criteria:

* the usual exclusion criteria for surgical techniques, pregnant patients, patiens under 18 patients who did not sign the informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To assess the tolerability of the laser diode in the treatment of endometrial polyps using a validated visual analogue pain scale | we we measure pain after resection of endometrial polyps, with 5 minutes for the patient thinks

SECONDARY OUTCOMES:
Determine if complete resection of polyps is achieved with both methods. | the duration of the polyp resection, subsequent assessment of the patient and her general condition. Time is measured, between 15 to 30 minutes
Compare the time spent on the removal of the polyp. | the duration of the polyp resection, subsequent assessment of the patient and her general condition. Time is measured, between 15 to 30 minutes
To evaluate the safety of both methods | the duration of the polyp resection, subsequent assessment of the patient and her general condition. Time is measured, between 15 to 30 minutes

OTHER OUTCOMES:
Assess the recurrence of polyps after 3 months of resection (another hysteroscopy). | 3 months after resection of the polyp, repeat hysteroscopy to assess recurrence, in 10 to 15 minutes. the patient is satisfied if foretaste and whether they would recommend the procedure.
Compare the degree of patient satisfaction with the different methods | 3 months after resection of the polyp, repeat hysteroscopy to assess recurrence, in 10 to 15 minutes. the patient is satisfied if foretaste and whether they would recommend the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: José Eduardo Arjona Berral, Gynecologist, Study Director — Head of the Department of Obstetrics and Gynecology at the University Hospital Reina Sofia; Maria Dolores Lara, Gynecologist, Principal Investigator — Physician specializing in obstetrics and gynecology.; Rafaela Dios Palomares, Engineer, Study Chair — Universidad de Córdoba
Locations (2):
- Spain (2):
  - Reina Sofia University Hospital, Córdoba, Cordoba
  - Reina Sofía University Hospital, Córdoba, Cordoba

REFERENCES:
- See also: Reina Sofia University Hospital in Cordoba, Spain — http://www.juntadeandalucia.es/servicioandaluzdesalud/hrs3/index.php?id=investigacion